CLINICAL TRIAL: NCT00132613
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Intra-pericardial Instillation of a Sclerosing Agent After Pericardial Drainage in Patients With Malignant Pericardial Effusion Associated With Lung Cancer (JCOG9811)
Brief Title: Trial of Drainage With or Without Bleomycin Instillation for Malignant Pericardial Effusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Tomohide Tamura , MD, Japan Clinical Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9811; C000000030
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Malignant Pericardial Effusion
Keywords: pulmonary neoplasm; malignant pericardial effusion; pericardial drainage; randomized trial; bleomycin; intrapericardial instillation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Procedure/Surgery: Observation alone after pericardial drainage
  Interventions: Procedure: Observation alone after pericardial drainage
- 2 (Experimental): Drug: Pericardial instillation of bleomycin after drainage
  Interventions: Drug: Pericardial instillation of bleomycin after drainage

INTERVENTIONS:
Procedure: Observation alone after pericardial drainage
  Arms: 1
Drug: Pericardial instillation of bleomycin after drainage
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of pericardial instillation of bleomycin as a sclerosing agent after pericardial drainage for lung cancer-associated malignant pericardial effusion.

DETAILED DESCRIPTION:
Malignant pericardial effusions (MPEs), which are commonly associated with cardiac tamponade, make oncologic emergencies requiring prompt drainage. In lung cancer patients, MPE is one of the most unpleasant terminal events. Drainage usually results in prompt palliation of symptoms, but recurrent effusions often occur. Sclerosis with pericardial instillation of various agents is reported to prevent the recurrence, and bleomycin is the most commonly used drug, with fewer toxicities compared with others. There is, however, no prospective trial of pericardial sclerosis as compared with drainage alone for MPEs, and it is far from clear whether sclerosis really benefits these patients in terminal stages.

Comparison: Intra-pericardial instillation of bleomycin after pericardial drainage versus drainage alone for MPEs caused by lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented lung cancer
* Clinically stable condition after pericardial drainage for malignant pericardial effusion (not necessary that it be documented by cytology)
* Expected to live 6 weeks or longer
* Sufficient organ function
* Signed informed consent

Exclusion Criteria:

* Myocardial infarction or unstable angina within 3 months
* Constrictive pericarditis
* Active pneumonitis
* Severe infection or disseminated intravascular coagulation (DIC)
* Other severe co-morbidity which could not be relieved with pericardial drainage
* Chemotherapy-naive small cell lung cancer

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 1999-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Survival without pericardial effusion at 2 months

SECONDARY OUTCOMES:
Successful extubation of pericardial drainage tube
time to extubation
survival without pericardial effusion at 1, 2, 4, 6, 12 months
symptom palliation
complication
long-term (> 6 months) effect on cardiac function

CONTACTS AND LOCATIONS:
Overall Officials: Tomohide Tamura, MD, Study Chair — National Cancer Center Hospital
Locations (31):
- Japan (31):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Aichi Cancer Center,Aichi Hospital, Okazaki,Kake-machi,Kuriyado,18, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Kyushu University Hospital, Fukuoka,Higashi-ku,Maidashi,3-1-1, Fukuoka
  - Gifu Municipal Hospital, Gifu,Kashima-cho,7-1, Gifu
  - Gunma Prefectural Cancer Center, Ota,Takabayashi-nishi-cho,617-1, Gunma
  - National Nishigunma Hospital, Shibukawa,Kanai,2854, Gunma
  - National Hospital Organization, Dohoku National Hospital, Asahikawa,Hanasaki,7-4048, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo,Shiroishi-ku,Kikusui,4-2-3-54, Hokkaido
  - Kobe City General Hospital, Kobe,Chuo-ku,Minatojimanakamachi,4-6, Hyōgo
  - Hyogo College of Medicine, Nishinomiya,Mukogawa-cho,1-1, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, Nishi-ibarakigun,Tomobemachi,Koibuchi,6528, Ibaraki
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Yokohama Mucipical Citizen's Hospital, Yokohama,Hodogaya-ku,Okazawa-cho,56, Kanagawa
  - Kumamoto Regional Medical Center Hospital, Kumamoto,Honjo,5-16-10, Kumamoto
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Osaka Prefectural Medical Center for Respiratory and Allergic Disease, Habikino,Habikino,3-7-1, Osaka
  - Rinku General Medical Center, Izumisano,rinku-ohrai-kita,2-23, Osaka
  - Graduate School of Medicine, Osaka City University, Osaka,Abeno-ku,Asahi-machi,1-5-7, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Kinki University School of Medicine, Osaka-Sayama,Ohno-higashi,377-2, Osaka
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai,Nagasone,1180, Osaka
  - National Hospital Organization Toneyama National Hospital, Toyonaka,Toneyama,5-1-1, Osaka
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - National Cancer Center Hospital, Chuo-ku,Tsukiji, 5-1-1, Tokyo
  - Cancer Institute Hospital, Koto-ku,Ariake,3-10-6, Tokyo
  - International Medical Center of Japan, Shinjuku-ku,Toyama,1-21-1, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata,Aoyagi,1800, Yamagata

REFERENCES:
- See also: Related Info — http://www.jcog.jp/